CLINICAL TRIAL: NCT03183986
Title: Comparison of the Efficacy of Phototherapy With Wavelength 478 vs. 459 nm for Treatment of Neonatal Jaundice Using Blue LED's.
Brief Title: Comparison of the Efficacy of Phototherapy Using Blue LED's With Wavelength 478 vs. 459 nm.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Pernille Kure Vandborg, Principal investigator, MD, PhD., University of Aarhus
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N-20160071
Record Dates: First submitted 2017-06-09; First posted 2017-06-12 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Neonatal Jaundice
MeSH Terms: conditions — Jaundice, Neonatal | interventions — Phototherapy

STUDY DESIGN:
Intervention Model Description: Infants are randomised to phototherapy with blue LED's with wavelength of 478 or 459 nm. The decrease of TSB between the groups is compared.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phototherapy 478 nm (Active Comparator): The jaundiced neonates receives phototherapy with blue light from above at wavelength 478 nm. They are treated for 24 hours, which is standard treatment for neonatal jaundice.
  Interventions: Device: Phototherapy
- Phototherapy 459 nm (Active Comparator): The jaundiced neonates receives phototherapy with blue light from above at wavelength 459 nm. They are treated for 24 hours, which is standard treatment for neonatal jaundice.
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy — Phototherapy for 24 hours.

SUMMARY:
Treatment of neonatal jaundice is phototherapy with blue light at wavelength about 460 nm and irradiance > 30 uw/cm2/nm. Though, recent in vitro models have suggested that a wavelength of 478 nm should be optimal in reducing total serum bilirubin. The aim of this study is therefore to compare the efficiency of phototherapy with light emitting diodes (LED's) of 478 vs. 459 nm., respectively.

DETAILED DESCRIPTION:
This is a prospective randomised study of the efficacy of phototherapy. Inclusion criteria are gestational age > 33 weeks and birth weight > 1800 grams, uncomplicated neonatal jaundice. The infants should be treated with phototherapy in a cradle for 24 hours, which is routine standard of care. Exclusion criteria is haemolytic disease. Total serum bilirubin (TSB) is measured before and after 24 hours of phototherapy. The infants are enrolled and randomised consecutively by the neonatologist using sealed and opaque envelopes.

Power calculation based on expected difference in decrease of TSB of 6% between the two groups and a significance level of 0.05, showed that 48 infants should be enrolled in each group.

ELIGIBILITY:
Inclusion Criteria:

* Indication for phototherapy with single light
* Gestational age > 33 weeks
* Birth weight > 1800 grams
* Should be treatable in a cradle

Exclusion Criteria:

* Haemolytic disease
* Indication for double/triple phototherapy or exchange transfusion

Ages: 25 Hours to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
Decrease of total serum bilirubin | 24 hours of phototherapy

CONTACTS AND LOCATIONS:
Overall Officials: Mette Donneborg, MD, Principal Investigator — Aalborg University Hospital
Locations (1):
- Neonatal department, Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lamola AA. A Pharmacologic View of Phototherapy. Clin Perinatol. 2016 Jun;43(2):259-76. doi: 10.1016/j.clp.2016.01.004. Epub 2016 Feb 15. PMID 27235206